CLINICAL TRIAL: NCT01882868
Title: A Single-Arm Phase II Study in Japan to Assess the Efficacy and Safety of Aflibercept Administered Every Two Weeks in Combination With FOLFIRI in Patients With Metastatic Colorectal Cancer Who Progressed During or Following an Oxaliplatin-Based Regimen
Brief Title: A Study of Aflibercept in Combination With FOLFIRI in Patients With Second-Line Metastatic Colorectal Cancer in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC11885; U1111-1120-0173 (Other: UTN)
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2016-08

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — aflibercept; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept + FOLFIRI (Experimental): Aflibercept 4 mg/kg intravenous (IV) infusion (1-2 hours) on Day 1 of Cycle 1 and every 2 weeks (q2w) thereafter, in combination with FOLFIRI regimen on Days 1-3 of Cycle 1 and q2w thereafter until disease progression (DP), unacceptable toxicity or participant's refusal. FOLFIRI regimen: IV infusions of levofolinate 200 mg/m^2 (2 hours) and irinotecan 180 mg/m^2 (90 minutes) simultaneously, followed by 5-FU 400 mg/m^2 IV bolus injection followed by continuous IV infusion of 5-FU (46 hours) at 2400 mg/m^2.
  Interventions: Drug: Aflibercept; Drug: Levofolinate; Drug: Irinotecan; Drug: 5-FU

INTERVENTIONS:
Drug: Aflibercept — Pharmaceutical form: Concentrated solution (100 mg/4 mL [25 mg/mL], 200 mg/8 mL [25 mg/mL]) for infusion; Route of administration: Intravenous
  Other Names: AVE0005
Drug: Levofolinate — Pharmaceutical form: Solution for infusion (marketed formulation); Route of administration: Intravenous
Drug: Irinotecan — Pharmaceutical form: Solution for infusion (marketed formulation); Route of administration: Intravenous
Drug: 5-FU — Pharmaceutical form: Solution for infusion (marketed formulation); Route of administration: Intravenous

SUMMARY:
Primary Objective:

To assess efficacy aflibercept + 5-fluorouracil (5-FU)/levofolinate/irinotecan (FOLFIRI) by objective response rate (ORR).

Secondary Objective:

To assess the following:

* safety profile;
* progression free survival (PFS);
* overall survival (OS);
* pharmacokinetics (PK);
* immunogenicity.

DETAILED DESCRIPTION:
Screening was up to 24 days. Treatment period was continued until DP, unacceptable toxicity, or participant's refusal. Follow up period was continued until death, participant's refusal, or end of study, whichever came first.

This trial was conducted in Japan, where the International Nonproprietary Name (INN) designation for the study molecule is "aflibercept" and this term is therefore used throughout the synopsis. In the US, the US proper name is "ziv-aflibercept".

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically proven adenocarcinoma of the colon or rectum.
* Metastatic disease that was not amenable to potentially curative treatment.
* Participants with measurable disease.
* One prior chemotherapeutic regimen (containing oxaliplatin) for metastatic disease.
* Participants who relapsed within 6 months of completion of oxaliplatin-based adjuvant chemotherapy were also eligible.

Exclusion criteria:

* Prior therapy with irinotecan.
* Less than 28 days elapsed from prior radiotherapy, prior surgery, or prior chemotherapy to the time of registration.
* Unresolved toxicity (grade >1) from prior anticancer therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status >1.
* Brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis.
* Other prior malignancy.
* Pregnant or breast-feeding women.
* Uncontrolled hypertension.
* Inadequate bone marrow function, liver function, or renal function.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (19):
- Japan (19):
  - Investigational Site Number 392011, Chiba
  - Investigational Site Number 392018, Chūōku
  - Investigational Site Number 392016, Fukuoka
  - Investigational Site Number 392017, Fukuoka
  - Investigational Site Number 392001, Kashiwa-Shi
  - Investigational Site Number 392019, Kawasaki-Shi
  - Investigational Site Number 392015, Matsuyama
  - Investigational Site Number 392013, Mitaka-Shi
  - Investigational Site Number 392004, Nagoya
  - Investigational Site Number 392006, Osaka
  - Investigational Site Number 392014, Sagamihara-Shi
  - Investigational Site Number 392008, Sapporo
  - Investigational Site Number 392003, Sendai
  - Investigational Site Number 392009, Shimotsuke-Shi
  - Investigational Site Number 392012, Shinjuku-Ku
  - Investigational Site Number 392005, Suita-Shi
  - Investigational Site Number 392002, Sunto-Gun
  - Investigational Site Number 392010, Tsukuba
  - Investigational Site Number 392007, Yufu-Shi

REFERENCES:
- [Derived] Hamaguchi T, Denda T, Kudo T, Sugimoto N, Ura T, Yamazaki K, Fujii H, Kajiwara T, Nakajima TE, Takahashi S, Otsu S, Komatsu Y, Nagashima F, Moriwaki T, Esaki T, Sato T, Itabashi M, Oki E, Sasaki T, Chiron M, Yoshino T. Exploration of potential prognostic biomarkers in aflibercept plus FOLFIRI in Japanese patients with metastatic colorectal cancer. Cancer Sci. 2019 Nov;110(11):3565-3572. doi: 10.1111/cas.14198. Epub 2019 Oct 21. PMID 31520559
- [Derived] Denda T, Sakai D, Hamaguchi T, Sugimoto N, Ura T, Yamazaki K, Fujii H, Kajiwara T, Nakajima TE, Takahashi S, Otsu S, Komatsu Y, Nagashima F, Moriwaki T, Esaki T, Sato T, Itabashi M, Oki E, Sasaki T, Sunaga Y, Ziti-Ljajic S, Brillac C, Yoshino T. Phase II trial of aflibercept with FOLFIRI as a second-line treatment for Japanese patients with metastatic colorectal cancer. Cancer Sci. 2019 Mar;110(3):1032-1043. doi: 10.1111/cas.13943. Epub 2019 Feb 22. PMID 30657223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 sites in Japan. A total of 68 participants were screened between 30 July 2013 and 12 March 2014, out of which 62 were enrolled and treated.
Pre-assignment Details: Among 68 participants screened, 6 were screen failures due to elevated urine protein-creatinine ratio (UPCR) and inadequate liver function tests (LFTs).
Period: Overall Study
Arm/Group | Aflibercept + FOLFIRI
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Evaluable participant (EP) population: all registered participants with measurable disease at study entry & with at least 1 valid post-baseline tumor evaluation. Participants who died due to DP or had documented radiological progressive disease before first post-baseline imaging evaluation were also included.
Groups:
- Aflibercept + FOLFIRI: Aflibercept 4 mg/kg IV infusion (1-2 hours) on Day 1 of Cycle 1 and q2w thereafter, in combination with FOLFIRI regimen on Days 1-3 of Cycle 1 and q2w thereafter until DP, unacceptable toxicity or participant's refusal. FOLFIRI regimen: IV infusions of levofolinate 200 mg/m^2 (2 hours) and irinotecan 180 mg/m^2 (90 minutes) simultaneously, followed by 5-FU 400 mg/m^2 IV bolus injection followed by continuous IV infusion of 5-FU (46 hours) at 2400 mg/m^2.
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 34
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Number; unit: participants] — ECOG PS is used to assess how the disease affects the daily living abilities of the participant. It ranges on the scale from 0-5 (0= normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead.
  participants
    0 | 40
    1 | 20
Prior Treatment with Bevacizumab [Number; unit: participants]
  Had Prior Treatment | 50
  Did Not Have Prior Treatment | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response
Description: Overall response in participants was defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) assessed by an independent radiological review committee (IRRC) according to response evaluation criteria in solid tumors (RECIST) version 1.1. CR was defined as disappearance of all target lesions; any lymph node (target or non-target) must have reduction in the short axis to <10 mm; PR was defined as at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. Percentage of participants with overall response and the 95% confidence interval (CI) were provided. The 95% CI was calculated using normal approximation.
Time Frame: Baseline and every 6 weeks until DP (maximum duration: 16.4 months)
Population: EP population: all registered participants with measurable disease at study entry & with at least 1 valid post-baseline tumor evaluation. Participants who died due to DP or had documented radiological progressive disease before first post-baseline imaging evaluation were also included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 60
percentage of participants | 8.3 [1.3 to 15.3]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval from the date of first study drug administration to the date of first observation of DP or death due to any cause, whichever came first. If death or progression was not observed, the participant was censored at the date of participant's last valid progression-free tumor assessment prior to the study cut-off date. DP for PFS was assessed by the IRRC based on tumor imaging according to RECIST 1.1. Progression in disease was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study with absolute increase of at least 5 mm, progression of existing non-target lesions, or presence of new lesions. PFS was estimated by Kaplan-Meier estimates.
Time Frame: Baseline and every 6 weeks until DP or death, due to any cause (maximum duration: 16.4 months)
Population: The safety population (all treated [AT] population) included all registered participants who received at least 1 (even if incomplete) infusion of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
months | 5.42 [4.140 to 6.702]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from the date of first study drug administration to the date of death due to any cause. If death was not observed, the participant was censored at the last date the participant was known to be alive or the study cut-off date, whichever was first. OS was estimated by Kaplan-Meier estimates.
Time Frame: Baseline up to death or study cut--off (maximum duration: 24.7 months)
Population: The safety population (AT population) included all registered participants who received at least 1 (even if incomplete) infusion of study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
months | 15.59 [11.203 to 19.811]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. TEAEs were defined as AEs that developed or worsened during the on--treatment period which was defined as the period from the time of first dose of study treatment until 30 days after the last dose of study treatment.
Time Frame: First dose (Day 1 of Cycle 1) of study treatment up to end of treatment visit (30 days after last dose of study treatment) (maximum duration: 77 weeks)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
participants | 62

5. Secondary Outcome: Aflibercept Immunogenicity Assessment: Number of Participants With Positive Sample(s) in the Anti-drug Antibodies (ADA) Assay and in the Neutralizing Anti-drug Antibodies (NAb) Assay
Description: Blood samples of participants were analyzed by using a titer-based, bridging immunoassay developed and validated to detect aflibercept ADA in human serum. Samples with positive antibody levels were further analyzed using a validated, non-quantitative, competitive ligand binding assay to detect NAb.
Time Frame: Baseline, at any time post baseline and 90 days after the last dose of aflibercept
Population: The safety population (AT population) included all registered participants who received at least 1 (even if incomplete) infusion of study treatment. Here 'n' signifies number of participants with available data for specified category.
Measure: Number; unit: participants
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
participants
  At baseline in the ADA assay (n=62) | 1
  At any time post-baseline in the ADA assay (n=62) | 0
  At any time post-baseline in the NAb assay (n=62) | 0
  At 90 days after last dose in the ADA assay (n=50) | 0
  At 90 days after last dose in NAb assay (n=50) | 0

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Free Aflibercept: ITT Population
Description: Sparse blood sampling was performed on 52 participants and additional blood sampling for detailed pharmacokinetic (PK) analysis was performed on 10 participants as per protocol. A population PK analysis was performed and an overall data is reported for all the participants.
Time Frame: Pre-dose, 1, 4, 24, 336 hours post aflibercept infusion on Day 1 of Cycle 1 for participants with sparse sampling & pre-dose, 1, 2, 4, 8, 24, 48, 168, 336 hours post aflibercept infusion on Day 1 of Cycle 1 for participants with additional sampling
Population: Intent-to-Treat (ITT) population included all registered participants.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
mcg/mL | 73.19 (10.72)

7. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to 14 Days Post Start of Infusion (AUC0-14 Day) for Free Aflibercept: ITT Population
Description: Sparse blood sampling was performed on 52 participants and additional blood sampling for detailed PK analysis was performed on 10 participants as per protocol. A population PK analysis was performed and an overall data is reported for all the participants.
Time Frame: as for outcome 6
Population: ITT population included all registered participants.
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
mcg*day/mL | 246.9 (41.1)

8. Secondary Outcome: Area Under the Concentration Time Curve (AUC) for Free Aflibercept: ITT Population
Description: as for outcome 7
Time Frame: as for outcome 6
Population: ITT population included all registered participants.
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
mcg*day/mL | 304.6 (62.8)

9. Secondary Outcome: Total Body Clearance (CL) for Free Aflibercept: ITT Population
Description: as for outcome 7
Time Frame: as for outcome 6
Population: ITT population included all registered participants.
Measure: Mean (Standard Deviation); unit: liter/day
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
liter/day | 0.8053 (0.1784)

10. Secondary Outcome: Volume of Distribution at the Steady State (Vss) for Free Aflibercept: ITT Population
Description: as for outcome 7
Time Frame: as for outcome 6
Population: ITT population included all registered participants.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 62
liters | 6.197 (1.106)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Free and Vascular Endothelial Growth Factor (VEGF)-Bound Aflibercept: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: In 10 participants of ITT population, additional blood samples were obtained for detailed non-compartmental PK analysis of free and VEGF-bound aflibercept in combination with irinotecan and 5-FU in Cycle 1.
Time Frame: Predose (prior to aflibercept infusion), 1, 2, 4, 8, 24, 48, 168 and 336 hours post aflibercept infusion on Day 1 of Cycle 1
Population: Subset of ITT population with additional blood sampling for detailed non-compartmental PK analysis. Number of participants analyzed=participants with PK assessment for the subset analysis. Here 'n' signifies number of participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
mcg/mL
  Plasma Free-Aflibercept (n=10) | 90.8 (16.5)
  Plasma VEGF-Bound Aflibercept (n=8) | 2.83 (0.836)

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration Observed (Tmax) for Free and VEGF-Bound Aflibercept in Cycle 1: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
days
  Plasma Free-Aflibercept (n=10) | 0.07 [0.04 to 0.09]
  Plasma VEGF-Bound Aflibercept (n=8) | 13.97 [7.01 to 16.05]

13. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUClast) for Free and VEGF-Bound Aflibercept: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
mcg*day/mL
  Plasma Free-Aflibercept (n=10) | 321 (58.9)
  Plasma VEGF-Bound Aflibercept (n=8) | 24.4 (6.17)

14. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to 14 Days Post Start of Infusion (AUC0-14 Day) for Free and VEGF-Bound Aflibercept: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
mcg*day/mL
  Plasma Free-Aflibercept (n=10) | 312 (51.8)
  Plasma VEGF-Bound Aflibercept (n=5) | 23.3 (2.45)

15. Secondary Outcome: Area Under the Concentration Time Curve (AUC) for Free Aflibercept: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: In 10 participants of ITT population, additional blood samples were obtained for detailed non-compartmental PK analysis of free aflibercept in combination with irinotecan and 5-FU in Cycle 1.
Time Frame: Pre-dose (prior to aflibercept infusion), 1, 2, 4, 8, 24, 48, 168 and 336 hours post aflibercept infusion on Day 1 of Cycle 1
Population: Subset of ITT population with additional blood sampling for detailed non-compartmental PK analysis. Number of participants analyzed=participants with PK assessment for the subset analysis.
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
mcg*day/mL | 355 (61.5)

16. Secondary Outcome: Total Body Clearance (CL) for Free Aflibercept: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 15
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter/day
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
liter/day | 0.716 (0.204)

17. Secondary Outcome: Volume of Distribution at the Steady State (Vss) for Free Aflibercept: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 15
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
liters | 3.53 (1.11)

18. Secondary Outcome: Terminal Elimination Half-life (t1/2z) for Free Aflibercept: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 15
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
days | 4.47 (0.680)

19. Secondary Outcome: Steady State Drug Concentration (Css) for 5-FU: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: In 10 participants of ITT population, additional blood samples were obtained for detailed non-compartmental PK analysis of 5-FU in combination with aflibercept and irinotecan in Cycle 1.
Time Frame: Pre-dose (prior to aflibercept infusion), 2.5, 21 and 45 hours post 5-FU infusion on Day 1 of Cycle 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
ng/mL | 930 (461)

20. Secondary Outcome: Clearance at Steady State (CLss) for 5-FU: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 19
Time Frame: Pre-dose (prior to aflibercept infusion), 2.5, 21 and 45 hours post 5-FU infusion on Day 1 of Cycle 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
liter/hour | 122 (76.2)

21. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Irinotecan and Its Active Metabolite SN-38: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: In 10 participants of ITT population, additional blood samples were obtained for detailed non-compartmental PK analysis of irinotecan and SN-38 in combination with aflibercept and 5-FU in Cycle 1.
Time Frame: Predose (prior to aflibercept infusion), 1.5, 2, 4.5 and 23 hours post irinotecan infusion on Day 1 of Cycle 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
ng/mL
  Plasma Irinotecan | 2220 (528)
  Plasma SN-38 | 32.2 (11.4)

22. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUClast) for Irinotecan and Its Active Metabolite SN-38: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 21
Time Frame: Pre-dose (prior to aflibercept infusion), 1.5, 2, 4.5 and 23 hours post irinotecan infusion on Day 1 of Cycle 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
ng*h/mL
  Plasma Irinotecan | 16900 (5970)
  Plasma SN-38 | 344 (173)

23. Secondary Outcome: Area Under the Concentration Time Curve (AUC) for Irinotecan and Its Active Metabolite SN-38: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 21
Time Frame: Pre-dose (prior to aflibercept infusion), 1.5, 2, 4.5 and 23 hours post irinotecan infusion on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
ng*h/mL
  Plasma Irinotecan (n=10) | 17700 (6400)
  Plasma SN-38 (n=4) | 341 (72.4)

24. Secondary Outcome: Terminal Elimination Half-life (t1/2z) for Irinotecan and Its Active Metabolite SN-38: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 21
Time Frame: Pre-dose (prior to aflibercept infusion), 1.5, 2, 4.5 and 23 hours post irinotecan infusion on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
hours
  Plasma Irinotecan (n=10) | 5.19 (0.736)
  Plasma SN-38 (n=5) | 10.3 (3.08)

25. Secondary Outcome: Active Metabolite SN-38 / Irinotecan Ratio on Area Under the Concentration Time Curve (Rmet): Participants With Additional Blood Sampling for Detailed PK Analysis
Description: In 10 participants of ITT population, additional blood samples were obtained for detailed non - compartmental PK analysis of irinotecan and SN-38 in combination with aflibercept and 5-FU in Cycle 1.
Time Frame: Pre-dose (prior to aflibercept infusion), 1.5, 2, 4.5 and 23 hours post irinotecan infusion on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
ratio | 0.0313 (0.0133)

26. Secondary Outcome: Total Body Clearance (CL) for Irinotecan: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: In 10 participants of ITT population, additional blood samples were obtained for detailed non-compartmental PK analysis of irinotecan in combination with aflibercept and 5-FU in Cycle 1.
Time Frame: Pre-dose (prior to aflibercept infusion), 1.5, 2, 4.5 and 23 hours post irinotecan infusion on Day 1 of Cycle 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
liter/hour | 18.3 (6.04)

27. Secondary Outcome: Volume of Distribution at the Steady State (Vss) for Irinotecan: Participants With Additional Blood Sampling for Detailed PK Analysis
Description: as for outcome 26
Time Frame: Predose (prior to aflibercept infusion), 1.5, 2, 4.5 and 23 hours post irinotecan infusion on Day 1 of Cycle 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Aflibercept + FOLFIRI
Number analyzed (Participants) | 10
liter | 92.5 (33.8)

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to the final visit (77 weeks) regardless of seriousness or relationship to investigational medicinal product.
Description: Reported AEs are TEAEs that is AEs that developed/worsened during the study treatment period (defined as the first study treatment administration to End-of-Treatment Visit [30 days of last infusion]).
Arm/Group | Aflibercept + FOLFIRI
Serious Adverse Events (participants affected / at risk) | 20/62
Other Adverse Events (participants affected / at risk) | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + FOLFIRI (N=62)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 4
Oesophagitis (Gastrointestinal disorders) | 1
Catheter site pain (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Biliary tract infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + FOLFIRI (N=62)
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 46
Abdominal pain (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 42
Nausea (Gastrointestinal disorders) | 36
Stomatitis (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 17
Fatigue (General disorders) | 38
Pyrexia (General disorders) | 13
Nasopharyngitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 4
Weight decreased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 46
Back pain (Musculoskeletal and connective tissue disorders) | 5
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 6
Proteinuria (Renal and urinary disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 30
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 7
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.